CLINICAL TRIAL: NCT04118231
Title: Comparison of the Effects of Dry Needling, Static Stretching and Instrument Assisted Soft Tissue Mobilization Techniques on Function, Performance and Muscle Structure in People With Hamstring Muscle Shortness
Brief Title: Effects of Dry Needling, Static Stretching and IASTM in People With Hamstring Muscle Shortness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, GÖKHAN MARAŞ, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019-114
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Hamstring Muscle Shortness and Elastographic Examination
Keywords: Hamstring Shortness; Dry Needling; Elastography
MeSH Terms: interventions — Dry Needling; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental)
  Interventions: Other: Dry needling
- Control group (No Intervention)

INTERVENTIONS:
Other: Dry needling — Group 1: Dry needling Group 2: static stretching Group 3: IASTM
  Other Names: IASTM, Static stretching
  Arms: Dry needling

SUMMARY:
The aim of this study was to investigate the effects of dry needling, static stretching and instrument assisted soft tissue mobilization on joint range of motion, performance and muscle structure in individuals with Hamstring muscle shortness and to examine the changes in soft tissue before and after application with the help of ultrasound elastography.

DETAILED DESCRIPTION:
The study was randomly divided into 3 groups. Group 1: Hamstring muscle group of patients for 5 minutes Instrument Assisted Soft Tissue Mobilization made of stainless steel instruments used by soft tissue mobilization by the therapist. In order to reduce friction and increase lubricity before application; If there is an unexpected erythema, edema or other unexpected side effects, the application will be stopped immediately.

2.Group: In the Hamstring muscle group of the patients, the acupuncture needles, which are made of stainless steel, sterile and disposable, will be applied under the supervision of an expert doctor for 30-45 seconds. In case of unexpected side effects, the application will be terminated.

Group 3: Patients' Hamstring muscle group under the supervision of the physiotherapist for a total of 5 minutes; A total of 10 repetitions of static tension will be applied for 30 seconds.

Before starting the study, anthropometric measurements, vertical and horizontal jump amounts of all participants will be measured before the application. Digital inclinometer will be used to determine the range of motion of the joint. Measurements will be made before and after the first application and the last measurement will be made 3 days after the end of 12 sessions. In addition, soft tissue changes in the hamstring muscle of the participants will be evaluated by US elastography before and at the end of the 12th session.

ELIGIBILITY:
Inclusion Criteria:

1. 18-35 age range
2. Volunteer to participate in the study
3. Not having a diagnosed condition

Exclusion Criteria:

1. Having any diagnosed discomfort
2. Being pregnant
3. Previously undergo surgery on the lower extremity
4. Physical therapy and rehabilitation of lower extremity in the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Range of motion | 4 weeks
  The amount of hip flexion will be measured using a digital inclinometer.
Muscle Strength | 4 weeks
  Muscle strength will be assessed in newton using a digital hand dinanometer.
Vertical jump | 4 weeks
  The amount of vertical jump will be calculated from the value of cm by the tape measure fixed to the wall.
Muscle stiffness | 4 weeks
  Muscle stiffness will be evaluated by an expert radiologist using ultrasound elastography.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Gökhan maraş, Ankara

IPD SHARING:
Plan to Share IPD: No